CLINICAL TRIAL: NCT05237063
Title: Prediction of Recurrence and Complications of Nephrolithiasis Using a Precision Medicine Approach
Acronym: PRECILITH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Institut Pasteur de Lille (Other); Université de Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2021_843_0137
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Kidney Stone; Nephrolithiasis
Keywords: Kidney Stone; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood and urine samples — Additional Blood and urine samples will be collected at inclusion, 1, 3 and 5 years follow up visits

SUMMARY:
Nephrolithiasis is a disease caused by the formation of kidney stones in the urinary tract which can then partially or completely obstruct the latter causing an extremely sharp pain called renal colic. In industrialized countries, it affects 10 to 20% of the population, and is the most common kidney disease.The primary objective of this study is to identify the clinical, biological, genetic, molecular and environmental determinants predictive of recurrence of renal lithiasis.

The study follow-up visit schedule corresponds to the visits usually scheduled as part of patient care: 1 year from the inclusion visit (A1), 3 years (A3) then 5 years (A5). Samples for research (additional volume of blood, urine) will be taken by a registered nurse along with the routine check-up samples.Samples intended for research will be sent by staff to the Biobanque de Picardie (CHU Amiens-Picardie) for processing and conservation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old), male or female ,
* Persons able to understand and object to the information provided (at the discretion of the investigator)
* Patient affiliated to social security
* Patient agreeing to sign the informed consent form
* patient having presented at least one renal colic attack before inclusion

Exclusion Criteria:

* Pregnant or breastfeeding woman.
* Persons deprived of liberty,
* Adults under legal protection guardianship, or curators or unable to express their consent.
* Patient refusing to participate in the study
* Patient in an emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with nephrolithiasis recurrence within 5 years of follow-up | at 5 years

SECONDARY OUTCOMES:
Occurrence of high blood pressure patients | at 1 year
Occurrence of high blood pressure patients | at 3 years
Occurrence of high blood pressure patients | at 5 years
Occurrence of patients with diabetes | at 1 year
Occurrence of patients with diabetes | at 3 year
Occurrence of patients with diabetes | at 5 year
Occurrence of patients with osteopenia | at 1 year
  Occurrence of patients with osteopenia during monitoring of bone mineral density with DXA
Occurrence of patients with osteopenia | at 3 year
  Occurrence of patients with osteopenia during monitoring of bone mineral density with DXA
Occurrence of patients with osteopenia | at 5 year
  Occurrence of patients with osteopenia during monitoring of bone mineral density with DXA
Occurrence of patients with a deterioration in renal function | at 1 year
  Occurrence of patients with a deterioration in renal function during follow-up
Occurrence of patients with a deterioration in renal function | at 3 year
  Occurrence of patients with a deterioration in renal function during follow-up
Occurrence of patients with a deterioration in renal function | at 5 year
  Occurrence of patients with a deterioration in renal function during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Nord, Amiens, France

IPD SHARING:
Plan to Share IPD: No